CLINICAL TRIAL: NCT03567928
Title: Anesthesiological Management of Ventilation With Laryngeal Mask in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) and Endoscopic Ultrasound Procedures
Brief Title: Laryngeal Mask in Upper Gastrointestinal Procedures
Acronym: SeoMask
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problem with device in study
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Agostoni Massimo, Principal Investigator, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43/int/2018
Record Dates: First submitted 2018-05-17; First posted 2018-06-26 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia; Airway Device; C.Surgical Procedure; Gastrointestinal
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Two groups: one receive sedation in spontaneous breathe, the other receive sedation with laryngeal mask
Who Masked: Participant
Masking Description: Induction of anesthesia and subsequent use (or not) of the device (laryngeal mask)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment (Active Comparator): Standard Treatment Sedation with propofol target controlled infusion (TCI) and no airway devices (mandatory spontaneous breathe)
  Interventions: Drug: Propofol
- Interventional Treatment (Experimental): Interventional Treatment Sedation with propofol target controlled infusion (TCI) and Gastro Cuff Pilot Laryngeal Mask (possibility to use a pressure-support ventilation)
  Interventions: Device: Sedation with Gastro Cuff Pilot Laryngeal Mask; Drug: Propofol

INTERVENTIONS:
Device: Sedation with Gastro Cuff Pilot Laryngeal Mask — This specific type of laryngeal mask allows to separate the gastric and respiratory tract and allows the anesthesiologist to support patient's ventilation as (and only if) necessary.
  Arms: Interventional Treatment
Drug: Propofol — Target controlled infusion (TCI) with propofol

SUMMARY:
Diagnostic and operative procedures of upper gastrointestinal (GI) tract are very common in all patients. Some procedures are difficult to tolerate because of long duration, prone position or significant stimulation of the upper airways. An example are endoscopic retrograde cholangiopancreatography (ERCP) and endoscopic pancreatic ultrasound.

The procedures are generally performed with deep sedation. Many pharmacologic regimens are available and described in literature. The investigator's institute adopts propofol target controlled infusion (TCI), which usually guarantees unconsciousness and unresponsiveness of patients. The main adverse event is dose-related respiratory depression. Pre-existing reasons for hypoventilation can exacerbate this event, especially in the elderly and the chronic obstructive pulmonary disease-patients. Laryngeal mask (LMA) is a useful tool to apply a pressure support ventilation. One specific type of LMA allows to separate the gastric and respiratory tract and, allows the anesthesiologist to support patient's ventilation as (and only if) necessary.

DETAILED DESCRIPTION:
This is a monocentric randomized controlled trial of superiority of LMA use in GI endoscopic procedures. Randomization is centralized. The study is single blind (patient). The study is no-profit. Every patients undergoing scheduled ERCP and endoscopic ultrasound will be screened and consecutive eligible patients will be enrolled. Subjects will be allocated according to a simple randomization list. The study starts after randomization and ends after discharge from the recovery room. After peripheral venous catheter insertion and vital parameters monitoring, patients will receive propofol TCI with a tailored target between 4 and 6 mcg/ml. The treatment group will receive LMA insertion and End-Tidal Carbon Dioxide (ETCO2) monitoring throughout the procedure. In case of hypoventilation, with an ETCO2 above 50 mmHg, the patient will be supported as necessary with PSV. The control group will not receive any airway device, according to the standard treatment. At the end of the procedure, both group will receive a laboratory testing (peripheral arterial sample), when the patient is still sedated. Vital parameters monitoring will continue in recovery room. Patients will be discharge as usual with an Aldrete score > 9.

Data will be collected during the procedure and in recovery room. Data will be stored in electronic database without mention to patient's name.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* written informed consent
* elective ERCP and endoscopic ultrasound procedure

Exclusion Criteria:

* pregnancy
* contraindication to propofol administration
* contraindication to mask insertion (e.g. malformation)
* emergency operation (not scheduled)
* preexisting causes of hypoventilation (e.g. chronic obstructive pulmonary disease, neuromuscular disease…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Partial Pressure of Carbon Dioxide (PaCO2) | Just before patient awakening (approximately 90-120 min after induction of anesthesia)
  PaCO2 level assessed by arterial sample

SECONDARY OUTCOMES:
Number of pressure support ventilation in treatment group | During the procedure
  Number needing pressure support ventilation (PSV) in the treatment group. A PSV will be performed in case of End-Tidal carbon dioxide level raising above 50 mmHg.
pH | Just before patient awakening (approximately 90-120 min after induction of anesthesia)
  pH assessed by arterial sample
Partial Pressure of Oxygen (PaO2) | Just before patient awakening (approximately 90-120 min after induction of anesthesia)
  PaO2 level assessed by arterial sample
Time to recover after the procedure | During recovery room stay (approximately 15-45 min after patient awakening)
  Time needed to recover: from arrival in recovery room to a Aldrete Score > 9
Satisfaction of the procedure operator | 1 minute after patient awakening
  Satisfaction of the operator assessed by a Likert 5 points-scale: 1 "Strongly disagree"; 2 "Disagree"; 3 " Neutral/Neither agree nor disagree"; 4 "Agree"; 5 "Strongly agree"
Satisfaction of the patient | 20 minutes after patient awakening
  Satisfaction of the patient assessed by a Likert 5 points-scale: 1 "Strongly disagree"; 2 "Disagree"; 3 " Neutral/Neither agree nor disagree"; 4 "Agree"; 5 "Strongly agree"
Number of completed endoscopic procedures | During the procedure
  Number of completed endoscopic procedures without necessity to change anesthesiological treatment or postpone the procedure for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Agostoni, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- San Raffaele Hospital, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03567928/Prot_SAP_000.pdf